CLINICAL TRIAL: NCT01248533
Title: Screening for Abdominal Aortic Aneurysm
Brief Title: Screening for Abdominal Aortic Aneurysm in 65 Year Old Males in Oslo
Acronym: AAAscreening
Status: Enrolling by invitation | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jorgen J Jorgensen, Professor dr.med., Oslo University Hospital
Other Study IDs: 2009/866
Record Dates: First submitted 2010-11-11; First posted 2010-11-25 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal aortic aneurysm, atherosclerosis
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Atherosclerosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Male subjects, 65 years of age, living in Oslo, Norway will be invited to be screened for abdominal aortic aneurysm.

DETAILED DESCRIPTION:
The invited population will be offered ultrasound investigation of their abdominal aorta. Further information regarding risk factors will be noted and measurement of ankle-brachial index will be measured/calculated. A further step in the future will be to sample blood with focus on different cytokines and genmediators.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 65 years

Exclusion Criteria:

* None

Ages: 65 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 65 year old males in Oslo
Sampling Method: Probability Sample
Enrollment: 7500 (Actual)
Dates: Start 2011-05; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Abdominal Aortic Aneurysm (AAA) | Yearly the number of patients with AAA among the screened population will be assessed during the inclusion period of 18 years..
  AAA definition: diameter equal or more than 30 mm. The number of identified patients with AAA will be yearlig assessed.

SECONDARY OUTCOMES:
Peripheral Arterial Disease (PAD) | Yearly the number of patients with PAD among the screened poplulation will be assessed during the inclusion period of 18 years.
  Investigate the prevalence of PAD among patients with AAA defined as having Ankle-Arm Index (AAI) less than 0.9. The number of these patients will be assessed yearly.

IPD SHARING:
Plan to Share IPD: Yes
All data are entered into the Electronic Patient Journal of Oslo University Hospital (DIPS)